CLINICAL TRIAL: NCT03399058
Title: A Randomized Cluster Controlled Study of an Interactive Voice Response Intervention and PD/Hearth ("PDH") to Improve Knowledge, Behavior Change, and Level of Confidence in Caregivers of Underweight Children in Cambodia
Brief Title: Innovative Nutrition and mHealth Evidence Building Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Public Health, Cambodia (Other Government)
Collaborators: World Vision International (Unknown); World Vision, Hong Kong (Unknown); World Vision, Cambodia (Unknown); Emory University (Other)
Responsible Party: Principal Investigator, ChheaChhorvann, Director of The National Institute of Public Health, National Institute of Public Health, Cambodia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 156NECHR
Record Dates: First submitted 2017-11-22; First posted 2018-01-16 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Underweight Children Aged 6-23 Month Old (WAZ < -1)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 5+5+5 (Control) (Other): The standard of care in Cambodia is known as the basic health and nutrition service package or 5+5+5. The participants in the first group will be the control group and will only be implementing the standard of care, 5+5+5 package (Group 1).
  Interventions: Other: Group 1 5+5+5 (Control)
- Group 2: 5+5+5 & PDH (Other): The participants in the second group will receive contextualized Hearth messages through on-going PDH programs in addition to the basic standard of care (Group 2). The Hearth messages are contextualized messages on child feeding practices that women in the community have found helpful to successfully prevent child malnutrition. This program will be delivered through in person community meetings.
  Interventions: Behavioral: Group 2: 5+5+5 & PDH
- Group 3: 5+5+5 & PDH lite+mHealth (Other): The participants in the third group will receive a similar program as group 2 with contextualized child feeding messages (PDH lite program) and receive follow-up through mobile support phone calls (Group 3).
  Interventions: Behavioral: Group 3: 5+5+5 & PDH lite+mHealth

INTERVENTIONS:
Other: Group 1 5+5+5 (Control) — The standard of care in Cambodia is known as the basic health and nutrition service package or 5+5+5. The participants in the first group will be the control group and will only be implementing the standard of care, 5+5+5 package (Group 1).
  Arms: Group 1 5+5+5 (Control)
Behavioral: Group 2: 5+5+5 & PDH — The participants in the second group will receive contextualized Hearth messages through on-going PDH programs in addition to the basic standard of care (Group 2).
  Arms: Group 2: 5+5+5 & PDH
Behavioral: Group 3: 5+5+5 & PDH lite+mHealth — The participants in the third group will receive a PDH lite program and receive follow-up through mobile support phone calls (Group 3).
  Arms: Group 3: 5+5+5 & PDH lite+mHealth

SUMMARY:
The project is the collaboration with the lead agencies National Institute of Public Health, World Vision and Emory University World Vision has a history of successfully implementing "Positive Deviance/Hearth (PDH)" programs across the globe. PDH is a community-based intervention utilizing locally appropriate health and infant feeding practices to rehabilitate underweight children and promote behavioral changes in caregivers. A recent systematic review on the PD/Hearth approach found that although some programs show clear success in particular settings, overall, the results were mixed for program effectiveness.

Furthermore, with the growing use of mobile phones and technology in the world, including Cambodia, there have been various studies and a systematic review that found SMS reminders and voice recordings to have promising impact on behavior change of patients for smoking cessation and improved adherence to drugs for asthma patients. Although there are positive findings around the use of mobile devices to improve behavior change, there has yet to be a study that examines the impact of mobile phones on improving behavior change of caregivers related to nutrition, water, sanitation and hygiene (WASH), health, and caring practices, which as a result, would decrease the prevalence of underweight in children 6-23 months of age.

This study will provide evidence on the effectiveness of the PDH model in Cambodia compared to the current standard of care. Investigators believe the PDH approach will be a powerful tool to reduce child malnutrition. In addition, given the intensity and cost burden associated with PDH, investigators will simultaneously test if the intensity of the PDH model can be reduced by introducing an innovative application of mHealth to replace 50% of face-to-face education sessions (5 days) and all follow up visits with mobile support calls. Collectively this research will provide critical data to inform program operations on the optimal and most effective method to reduce child underweight in Cambodia.

In Year 1, the purpose of this study is to assess the effectiveness of contextualized messages through PDH programs and a mobile technology (mHealth), to improve knowledge, behaviour change, and level of confidence of caregivers with underweight children aged 6-23 months in feeding, hygiene, health-seeking, and caring practices. In Year 2, the study's aim will be to assess the prevention of underweight in the siblings of the children included in the three programs outside of the 360 study subjects from Year 1.

ELIGIBILITY:
Inclusion Criteria for Enrollment:

* Child 6-23 months residing in study area and intending to stay in area for study duration
* Underweight child (Weight for Age Z-score < -1)

Exclusion Criteria:

* No access to mobile phone
* Severe Acute malnutrition (Weight for Height Z-score <-3), Edema

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in prevalence of underweight children over time | Measured at Baseline (Month 0), Midline (Month 3), Endline (Month 12)
  Weight, height/length and MUAC will be measured at Baseline (Month 0), Month 3, and Month 12. The data such as weight, height/length, MUAC, gender, and date of birth are needed to calculate the prevalence of underweight children. These data will be entered into the software ENA2015 to compare the weight-for-age, MUAC, height-for-age, and weight-for-height data to the international WHO reference standards in order to identify the underweight status of the children. The investigators will assess the difference in prevalence of underweight children among the three arms between baseline (Month 0), midline (month 3), and endline (month 12).
Change in mean of weight (grams) over time | Measured at Baseline (Month 0), Midline (Month 3), Endline (Month 12)
  Weight, height/length and MUAC will be measured at Baseline (month 0), Month 3, and Month 12. The investigators will assess the change in mean of weight (grams) among the three arms between baseline (Month 0), midline (month 3), and endline (month 12).
Change in percentage of caregivers correctly answering questions on child feeding, hygiene, health-seeking and caring practices over time | Measured at Baseline (Month 0), Midline (Month 3), Endline (Month 12)
  The investigators will assess the knowledge improvement regarding the child feeding, hygiene, health-seeking and caring practices between Baseline (Month 0), Midline (Month 3), Endline (Month 12) through quantitative questionnaire. The questionnaire was established by the research team which consists of topic around child feeding, hygiene, caring, health-seeking practices.
Change in percentage of caregivers who have adopted proper child feeding, hygiene, health-seeking, and caring practices | Measured at Baseline (Month 0), Midline (Month 3), Endline (Month 12)
  The investigators will assess the behavioral change regarding the child feeding, hygiene, health-seeking and caring practices between Baseline (Month 0), Midline (Month 3), Endline (Month 12) through quantitative questionnaire. The questionnaire was established by the research team which consists of topic around child feeding, hygiene, caring, health-seeking practices.
Change in percentage of caregivers self-reporting confidence in ability to adopt proper child feeding, hygiene, health-seeking, and caring practices over time | Measured at Baseline (Month 0), Midline (Month 3), Endline (Month 12)
  The investigators will assess the confident level in ability to adopt proper child feeding, hygiene, health-seeking, and caring practics between Baseline (Month 0), Midline (Month 3), Endline (Month 12) through quantitative questionnaire. The questionnaire was established by the research team which consists of topic around child feeding, hygiene, caring, health-seeking practices.
Assess the percentage of siblings of enrolled children in each group with a weight for height z-score <-2 | Measured at Year 2 Endline
  Assessment of the percentage of underweight younger siblings of the child who was admitted into the program will be assessed through rapid survey. Younger siblings of the enrolled children will be measured weight, height/length and MUAC at the Year 2 endline. The data such as weight, height/length, MUAC, gender, and date of birth are needed to calculate the prevalence of underweight children. These data will be entered into the software ENA2015 to compare the weight-for-age, MUAC, height-for-age, and weight-for-height data to the international WHO reference standards in order to identify the underweight status of the children. The investigators will assess the difference in prevalence of underweight children among the three arms.

CONTACTS AND LOCATIONS:
Locations (3):
- Cambodia (3):
  - ADP Samrong Tong 2, Kampong Speu, Kamong Speu
  - ADP Boribor 2, Kampong Chhnang
  - ADP Rolea Phaea, Kampong Chhnang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Baik D, Reinsma K, Chhorvann C, Oy S, Heang H, Young MF. Program Impact Pathway of the Positive Deviance/Hearth Interactive Voice Calling Program in a Peri-Urban Context of Cambodia. Curr Dev Nutr. 2022 Mar 28;6(5):nzac045. doi: 10.1093/cdn/nzac045. eCollection 2022 May. PMID 35611354